CLINICAL TRIAL: NCT03492749
Title: Busulfan Concentration in Saliva and Plasma, and Its Relationship With Salivary Changes and Mucositis in the Digestive Tract of Patients Submitted to Hematopoietic Stem Cell Transplantation
Status: Completed | Type: Observational
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Principal Investigator, Fernanda de Paula Eduardo, Dentist, Hospital Israelita Albert Einstein
Other Study IDs: 2902-16
Record Dates: First submitted 2018-04-02; First posted 2018-04-10 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Bone Marrow Disease
MeSH Terms: conditions — Bone Marrow Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group Busulfan: Patients submitted a Bone marrow transplantation with the busulfan chemotherapy in the conditioning. Saliva monitoring
  Interventions: Diagnostic Test: Saliva monitoring
- Group no busulfan: Patients submitted a Bone marrow transplantation without busulfan chemotherapy in the conditioning.Saliva monitoring
  Interventions: Diagnostic Test: Saliva monitoring

INTERVENTIONS:
Diagnostic Test: Saliva monitoring — The first objective of this project is to verify the feasibility of using the analysis of salivary concentration of BU during individual adjustments of this drug in the period that precedes HSCT

SUMMARY:
Busulfan (Bu) has been widely used for the treatment of neoplastic and non-neoplastic hematological disturbances, with satisfactory results in terms of successful hematopoietic stem cell transplantation (HSCT). Individual monitoring of the Bu dosage, which is done by means of various blood sample collections, is necessary for the purpose of attaining ideal therapeutic levels and minimizing systemic toxicity. This procedure sometimes becomes costly to and uncomfortable for the patient. Saliva has been analyzed as a possible alternative fluid for this monitoring.

DETAILED DESCRIPTION:
The first objective of this project is to verify the feasibility of using the analysis of salivary concentration of BU during individual adjustments of this drug in the period that precedes HSCT. Another question related to this project is with reference to the effects that the Bu concentration in saliva has on the mucosa of the digestive tract, particularly with regard to mucositis and salivary changes. Thus, the second objective of this project is to verify whether there is any association between salivary changes, cytological changes in the oral mucosa, degrees of mucositis and concentration of Bu in saliva. An analysis will be performed of the Bu concentration in saliva and in blood, as well as the salivary dosage of total proteins, albumin, amylase, antioxidant enzymes (superoxide dismutase, catalase, and glutathione reductase) and pro-inflammatory cytokines IL-1β, IL-6 and TNF-α. In addition, morphological analysis will be made, and rate of apoptosis of cells of the oral mucosa will be analyzed. If the efficacy of saliva for the individual adjustment of the dose of Bu is confirmed, this method could facilitate the dissemination of pharmacokinetic monitoring of this drug in chemotherapy and HSCT centers. In addition, it is expected that the results of the present project will allow establishment of the toxicity indicators of BU detected by analysis of saliva and the cells of the oral mucosa, thereby allowing the early adoption of preventive actions for reducing the frequency and severity of mucositis, a fact that may have a positive impact on the success of HSCT.

ELIGIBILITY:
Inclusion Criteria:

* Submitted a TCTH

Exclusion Criteria:

* No signed informed consent

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients submitted bone marrow transplantation
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
descriptive Analysis salivar | 2 years
  An analysis will be performed of the Bu concentration in saliva and in blood, as well as the salivary dosage of total proteins, albumin, amylase, antioxidant enzymes

IPD SHARING:
Plan to Share IPD: No